CLINICAL TRIAL: NCT02252445
Title: Effect of Propofol and Sevoflurane on Postoperative Catheter-Related Bladder Discomfort
Brief Title: Propofol and Sevoflurane for Catheter-Related Bladder Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRBDPPFSEVO
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2014-09

CONDITIONS: Catheter Site Discomfort; Complications; Anesthesia; Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): Propofol will be administered as the anesthetic maintenance agent.
  Interventions: Drug: Propofol
- Sevoflurane (Experimental): Sevoflurane will be administered as the anesthetic maintenance agent.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Propofol will be administered.
  Arms: Propofol
Drug: Sevoflurane — Sevoflurane will be administered.
  Arms: Sevoflurane

SUMMARY:
The investigators want to evaluate the efficacy of the propofol and sevoflurane for the prevention of catheter-related bladder discomfort.

DETAILED DESCRIPTION:
The mechanism of catheter-related bladder discomfort is thought to be related to the muscarinic receptor. Propofol and desflurane are most widely used as an anesthetic agent. Propofol and desflurane are known to block the muscarinic receptor in different ways.

The investigators want to evaluate the efficacy of the propofol and sevoflurane for the prevention of catheter-related bladder discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for transurethral bladder excision under general anesthesia
* ASA I-III

Exclusion Criteria:

* Foley catheter less than 18 Fr.
* Patients with obstruction of urinary tract
* Patients with neurogenic bladder
* Patients with severe obesity
* Patients with neurologic disorder
* Patients with chronic pain
* Patients with allergic history to propofol or sevoflurane

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seolu National University of Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol | Sevoflurane
Started | 41 | 41
Completed | 41 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Sevoflurane | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 22 | 22 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 32 | 30 | 62
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Catheter-related Bladder Discomfort
Description: Catheter-related bladder discomfort will be measured at 1 hour postoperatively (0:none, 1:mild, 2:moderate, 3:severe). Patients with score >0 will be counted.
Time Frame: 1 hour postoperatively
Population: Patients with score >0 were counted.
Measure: Number; unit: participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
participants | 35 | 24

2. Secondary Outcome: Catheter-related Bladder Discomfort
Description: as for outcome 1
Time Frame: 0, 6 and 24 hour postoperatively
Population: Patients with score >0 will be counted.
Measure: Number; unit: participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
participants | 38 | 27

3. Secondary Outcome: Hemodynamic Parameters
Description: Mean blood pressure and heart rate will be measured at 0, 1, 5, 10 minute postoperatively. Measurement at 10 minute means Mean blood pressure and heart rate at the admission of post-anesthetic care unit.
Time Frame: 0, 1, 5, 10 minute postoperatively
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
mmHg | 90 (24) | 88 (27)

4. Secondary Outcome: Nausea
Description: Nausea will be measured at 0, 1, 6 and 24 hour postoperatively.
Time Frame: 0, 1, 6 and 24 hour postoperatively
Population: Patients with nausea were counted.
Measure: Number; unit: participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
participants | 2 | 3

5. Secondary Outcome: Vomiting
Description: Vomiting will be measured at 0, 1, 6 and 24 hour postoperatively.
Time Frame: 0, 1, 6 and 24 hour postoperatively
Population: Patients with vomiting were counted.
Measure: Number; unit: participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
participants | 2 | 1

6. Secondary Outcome: Dry Mouth
Description: Dry mouth will be measured at 0, 1, 6 and 24 hour postoperatively.
Time Frame: 0, 1, 6 and 24 hour postoperatively
Population: Patients with dry mouth were counted.
Measure: Number; unit: participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
participants | 2 | 2

7. Secondary Outcome: Flushing
Description: Flushing will be measured at 0, 1, 6 and 24 hour postoperatively.
Time Frame: 0, 1, 6 and 24 hour postoperatively
Population: Patients with flushing were counted.
Measure: Number; unit: participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
participants | 0 | 0

8. Secondary Outcome: Blurred Vision
Description: Blurred vision will be measured at 0, 1, 6 and 24 hour postoperatively.
Time Frame: 0, 1, 6 and 24 hour postoperatively
Population: Patients with blurred vision were counted.
Measure: Number; unit: participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
participants | 0 | 0

9. Secondary Outcome: Dizziness
Description: Dizziness will be measured at 0, 1, 6 and 24 hour postoperatively.
Time Frame: 0, 1, 6 and 24 hour postoperatively
Population: Patients with dizziness were counted.
Measure: Number; unit: participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
participants | 0 | 0

10. Secondary Outcome: Analgesics
Description: The amount of analgesics will be measured at 0, 1, 6 and 24 hour postoperatively.
Time Frame: 0, 1, 6 and 24 hour postoperatively
Population: Patients infused with tramadol were counted.
Measure: Number; unit: participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 41 | 41
participants | 22 | 13

ADVERSE EVENTS:
Time Frame: 0 h, 1 h, 6 h, 24 h, 6 month
Arm/Group | Propofol | Sevoflurane
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes